CLINICAL TRIAL: NCT06070298
Title: Smartphone-Based Use of Phonocardiography Technique for Detection of Murmurs: Diagnostic Performance Study Protocol
Brief Title: Can a Smartphone Listen to Your Heart? A Performance Study on Detecting Abnormalities in Your Heart Sounds
Acronym: AUSC1
Status: Active, not recruiting | Type: Observational
Sponsor: Wong Chun Ka (Other)
Collaborators: Laboratory of Data Discovery for Health (Unknown); The University of Hong Kong (Other)
Responsible Party: Sponsor-Investigator, Wong Chun Ka, Clinical Assistant Professor, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Other Study IDs: AUSC1
Record Dates: First submitted 2023-09-29; First posted 2023-10-06 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Valvular Heart Disease; Heart Murmurs; Cardiovascular Abnormalities
Keywords: Auscultation; Smartphone; Heart Sounds; Heart Auscultation; Phonocardiography; Stethoscopes; Telemedicine
MeSH Terms: conditions — Heart Valve Diseases; Heart Murmurs; Cardiovascular Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Abnormal Echocardiography Diagnosis: Participants with abnormal echocardiography diagnosis within three years.
  Interventions: Diagnostic Test: Computer algorithms
- Normal Echocardiography Diagnosis: Participants with normal echocardiography diagnosis within three years.
  Interventions: Diagnostic Test: Computer algorithms

INTERVENTIONS:
Diagnostic Test: Computer algorithms — Collection of lightweight computer algorithms called ausculto™ that is designed to perform real-time heart sound analysis to detect heart murmur.
  Other Names: ausculto™; Vitogram™

SUMMARY:
This observational study aims to assess the performance of the software called ausculto™. ausculto™ is a collection of computer algorithms that intend to analyse heart sounds recorded from the built-in microphone of a smartphone for abnormal sounds.

Participants will have their heart sounds recorded during their regular clinic appointment after consenting to participate in this study.

Researchers will manually annotate the recorded heart sounds to create a database for use in future training and testing of artificial intelligence (AI) intended for medical uses.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥22 years (adult)
* Outpatients who have undergone echocardiography within 3 years at their normal non-research follow-up clinic visit appointment

Exclusion Criterion:

* Implanted active medical devices in the torso, such as pacemakers and defibrillators

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult hospital cardiology out-patients (22-year-old and above) who have undergone echocardiography within 3 years at their normal non-research follow-up clinic visit appointment.
Sampling Method: Non-Probability Sample
Enrollment: 577 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of ausculto™ Using Auscultation Paired with Echocardiography as Ground Truth | Day 0
  Sensitivity is defined as the percentage of true positives out of all positive cases from the ground truth. Cardiologist electronic stethoscope heart sound recording annotations paired with echocardiography diagnosis will be used as the ground truth. Heart sound recordings from electronic stethoscope will be rated by two independent cardiologists for presence or absence of murmur, with a third cardiologist consulted in case of disagreement.
Specificity of ausculto™ Using Auscultation Paired with Echocardiography as Ground Truth | Day 0
  Specificity is defined as the percentage of true negatives out of all negative cases from the ground truth. Cardiologist electronic stethoscope heart sound recording annotations paired with echocardiography diagnosis will be used as the ground truth. Heart sound recordings from electronic stethoscope will be rated by two independent cardiologists for presence or absence of murmur, with a third cardiologist consulted in case of disagreement.

SECONDARY OUTCOMES:
Sensitivity of ausculto™ Using Auscultation as Ground Truth | Day 0
  Sensitivity is defined as the percentage of true positives out of all positive cases from the ground truth. Cardiologist electronic stethoscope heart sound recording annotations will be used as the ground truth. Heart sound recordings from electronic stethoscope will be rated by two independent cardiologists for presence or absence of murmur, with a third cardiologist consulted in case of disagreement.
Specificity of ausculto™ Using Auscultation as Ground Truth | Day 0
  Specificity is defined as the percentage of true negatives out of all negative cases from the ground truth. Cardiologist electronic stethoscope heart sound recording annotations will be used as the ground truth. Heart sound recordings from electronic stethoscope will be rated by two independent cardiologists for presence or absence of murmur, with a third cardiologist consulted in case of disagreement.
Sensitivity of ausculto™ Using Echocardiography as Ground Truth | Day 0
  Sensitivity is defined as the percentage of true positives out of all positive cases from the ground truth. Echocardiography diagnosis will be used as the ground truth.
Specificity of ausculto™ Using Echocardiography as Ground Truth | Day 0
  Specificity is defined as the percentage of true negatives out of all negative cases from the ground truth. Echocardiography diagnosis will be used as the ground truth.
Positive Predictive Value of ausculto™ Using Auscultation Paired with Echocardiography as Ground Truth | Day 0
  Positive predictive value is defined as the percentage of true positives out of all positive results from ausculto™. Cardiologist electronic stethoscope heart sound recording annotations paired with echocardiography diagnosis will be used as the ground truth. Heart sound recordings from electronic stethoscope will be rated by two independent cardiologists for presence or absence of murmur, with a third cardiologist consulted in case of disagreement.
Negative Predictive Value of ausculto™ Using Auscultation Paired with Echocardiography as Ground Truth | Day 0
  Negative predictive value is defined as the percentage of true negatives out of all negative results from ausculto™. Cardiologist electronic stethoscope heart sound recording annotations paired with echocardiography diagnosis will be used as the ground truth. Heart sound recordings from electronic stethoscope will be rated by two independent cardiologists for presence or absence of murmur, with a third cardiologist consulted in case of disagreement.
Positive Predictive Value of ausculto™ Using Auscultation as Ground Truth | Day 0
  Positive predictive value is defined as the percentage of true positives out of all positive results from ausculto™. Cardiologist electronic stethoscope heart sound recording annotations will be used as the ground truth. Heart sound recordings from electronic stethoscope will be rated by two independent cardiologists for presence or absence of murmur, with a third cardiologist consulted in case of disagreement.
Negative Predictive Value of ausculto™ Using Auscultation as Ground Truth | Day 0
  Negative predictive value is defined as the percentage of true negatives out of all negative results from ausculto™. Cardiologist electronic stethoscope heart sound recording annotations will be used as the ground truth. Heart sound recordings from electronic stethoscope will be rated by two independent cardiologists for presence or absence of murmur, with a third cardiologist consulted in case of disagreement.
Positive Predictive Value of ausculto™ Using Echocardiography as Ground Truth | Day 0
  Positive predictive value is defined as the percentage of true positives out of all positive results from ausculto™. Echocardiography diagnosis will be used as the ground truth.
Negative Predictive Value of ausculto™ Using Echocardiography as Ground Truth | Day 0
  Negative predictive value is defined as the percentage of true negatives out of all negative results from ausculto™. Echocardiography diagnosis will be used as the ground truth.
Number of Adverse Events Reported by Participants Deemed to be Caused by the Observational Procedures | Day 0 to Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Chun Ka Wong, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong SAR, China

IPD SHARING:
Plan to Share IPD: No